CLINICAL TRIAL: NCT00857415
Title: A Phase III Study of the Correlation Between Florbetapir F 18 (18F-AV-45) PET Imaging and Amyloid Pathology
Brief Title: Phase III Study of the Correlation Between Florbetapir F18 PET Imaging and Amyloid Pathology in the Brain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A07
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
Keywords: florbetapir F 18 PET; amyloid imaging; Amyloid pathology in the brain
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autopsy Cohort (Experimental): End-of-life subjects (life expectancy < 6 months) consenting to brain donation at autopsy.
  Interventions: Drug: florbetapir F 18
- Specificity Cohort (Experimental): Younger healthy controls presumed to be devoid of beta-amyloid plaques.
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — Single i.v. bolus injection of 370MBq (10 mCi) followed by saline flush, 50 minutes prior to imaging, 10 minute image duration
  Other Names: 18F-AV-45; AV-45; Amyvid

SUMMARY:
The study is designed to test the relationship between measurements of brain amyloid using florbetapir F 18 PET imaging and true levels of amyloid by dissection of the brain at autopsy. Amyloid in the brain is a key feature of Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
There will be two primary analyses:

* The first primary analysis will evaluate the correlation between the blinded readers' rating of amyloid plaque density on the PET scan and the cortical amyloid plaque density at autopsy.
* The second primary analysis will evaluate the specificity of the blinded readers' rating of presence or absence of amyloid plaque density on the PET scan

For the autopsy population, subjects will be enrolled from various end-of-life (e.g. hospice / hospital / nursing home) and late-life (longitudinal studies of aging) populations. Enrollment will include subjects with various levels of cognitive status, ranging from cognitively normal through dementia. It is expected that amyloid plaque density in this elderly population will range from very low (normal aging) through moderate (e.g. cognitively normal subjects with asymptomatic amyloid deposits or mild cognitive impairment (MCI) subjects with intermediate levels of amyloid deposits) to very high (subjects with AD). The study will also enroll younger healthy subjects presumably devoid of amyloid in the specificity cohort.

Screening assessments may take place over several days and will include collection of demographic information, diagnostic interview, and safety assessments. At the time of screening, subjects or caregivers will be asked to provide consent for brain donation if they are not already enrolled in a brain donation program affiliated with this study, in addition to providing informed consent for the screening and imaging procedures in the study.

Subjects who qualify for the study will have a catheter placed for intravenous (i.v.) administration of florbetapir F 18. Subjects will receive a single i.v. bolus of 370 MBq (10 mCi) of florbetapir F 18 followed by brain PET imaging for 10 minutes duration, beginning approximately 50 minutes post-injection. Vital signs and safety labs will be obtained prior to the administration of florbetapir F 18 and at the completion of the imaging session. Adverse events will be continuously monitored during the imaging session. Subjects who experience an adverse event will not be discharged until the event has been resolved or stabilized.

ELIGIBILITY:
Inclusion Criteria (autopsy cohort):

* Have a projected life expectancy of ≤ 6 months as determined by the principal investigator (e.g. terminal medical condition) or are already enrolled in a longitudinal study of aging with an autopsy component;
* Can tolerate a 10 minute PET scan; and
* Give informed consent for study procedures and brain donation consistent with the legal requirements of the State in which they are enrolled and the State in which they die.

Inclusion Criteria (specificity cohort):

* Cognitively and neurologically healthy males and females 18 to 40 years of age;
* Who had no known risk factors for AD, including:
* Known genetic risk factors for AD, including an ApoE ε4 allele (note: ApoE genotype was determined after enrollment and was not disclosed to healthy control subjects). Scans from subjects carrying an ApoE ε4 allele were not included in the primary specificity analysis, but were included in an exploratory analysis;
* First degree relative with a known progressive dementing disorder;
* History of cognitive decline;
* History of neurologic, neurodegenerative, or psychiatric disease;
* History of head trauma; or
* Evidence of brain abnormality on a MRI scan;
* Who performed in an age-appropriate normal range on the Wechsler Logical Memory I & II, story A;
* Who could tolerate a 10-minute PET scan; and
* Who provided informed consent before any study procedures were performed.

Exclusion Criteria:

* Have primary brain tumor, known metastases to the brain, central nervous system (CNS) lymphoma;
* Have any major, focal structural loss of brain matter;
* Are aggressively being treated with life sustaining measures (e.g. currently on respirator; receiving high dose chemotherapy);
* Have a clinically significant infectious disease, including Acquired Immune Deficiency Syndrome (AIDS), Human Immunodeficiency Virus (HIV) infection, previous positive test for hepatitis or HIV or Creutzfeldt-Jakob disease (CJD);
* Are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days;
* Have ever participated in an experimental study with an amyloid targeting agent (e.g. anti-amyloid immunotherapy, secretase inhibitor);
* Have had a radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session; or
* Are females of childbearing potential who are pregnant or not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (25):
- United States (25):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Irvine, California
  - Research Site, San Francisco, California
  - Research Site, Fort Myers, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Hattiesburg, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Albany, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Durham, North Carolina
  - Research Site, Centerville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Charleston, South Carolina
  - Research Site, Johnson City, Tennessee
  - Research Site, Bennington, Vermont

REFERENCES:
- [Result] Clark CM, Schneider JA, Bedell BJ, Beach TG, Bilker WB, Mintun MA, Pontecorvo MJ, Hefti F, Carpenter AP, Flitter ML, Krautkramer MJ, Kung HF, Coleman RE, Doraiswamy PM, Fleisher AS, Sabbagh MN, Sadowsky CH, Reiman EP, Zehntner SP, Skovronsky DM; AV45-A07 Study Group. Use of florbetapir-PET for imaging beta-amyloid pathology. JAMA. 2011 Jan 19;305(3):275-83. doi: 10.1001/jama.2010.2008. PMID 21245183
- [Derived] Clark CM, Pontecorvo MJ, Beach TG, Bedell BJ, Coleman RE, Doraiswamy PM, Fleisher AS, Reiman EM, Sabbagh MN, Sadowsky CH, Schneider JA, Arora A, Carpenter AP, Flitter ML, Joshi AD, Krautkramer MJ, Lu M, Mintun MA, Skovronsky DM; AV-45-A16 Study Group. Cerebral PET with florbetapir compared with neuropathology at autopsy for detection of neuritic amyloid-beta plaques: a prospective cohort study. Lancet Neurol. 2012 Aug;11(8):669-78. doi: 10.1016/S1474-4422(12)70142-4. Epub 2012 Jun 28. Erratum In: Lancet Neurol. 2012 Aug;11(8):658. PMID 22749065

RESULTS

PARTICIPANT FLOW:
Groups:
- Autopsy Cohort: End-of-life subjects consenting to brain donation at autopsy. Subjects received a single intravenous injection of 370 MBq florbetapir followed by a 10-minute PET scan 50 minutes post-injection.
- Specificity Cohort: Younger healthy controls presumed to be devoid of beta-amyloid plaques. Subjects received a single intravenous injection of 370 MBq florbetapir followed by a 10-minute PET scan 50 minutes post-injection.
Period: Overall Study
Arm/Group | Autopsy Cohort | Specificity Cohort
Started | 152 | 74
Deceased Within One Year of AV-45 Scan | 37 | 0 (Subjects in the specificity cohort were not followed to autopsy)
Completed | 35 | 74
Not Completed | 117 | 0
Not completed — Image acquisition failure | 2 | 0
Not completed — Invalid image or not imaged | 3 | 0
Not completed — Subject still living at end of study | 110 | 0
Not completed — Deceased with no autopsy | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autopsy Cohort | Specificity Cohort | Total
Number analyzed (Participants) | 152 | 74 | 226
Age Continuous [Mean (Standard Deviation); unit: years] | 78.1 (13.35) | 26.6 (6.50) | 61.3 (26.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 26 | 107
  Male | 71 | 48 | 119
Region of Enrollment [Number; unit: participants]
  United States | 152 | 74 | 226

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Florbetapir-PET Image and Amyloid Plaque Density
Description: Spearman's rank order correlation of the median semi-quantitative visual read of the florbetapir-PET image and the amyloid plaque density assessed post-mortem by quantitative immunohistochemistry (IHC) averaged across 6 brain regions (precuneus, parietal cortex, frontal cortex, temporal cortex, posterior cingulate, anterior cingulate). Spearman's rank order correlation ranges from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: at autopsy up to 12 months post-scan
Population: All subjects with a valid image who came to autopsy within 1 year of scan, minus 6 subjects who served as front-runners
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Autopsy Cohort: End-of-life subjects consenting to brain donation at autopsy
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 29
Correlation coefficient | 0.78 [0.58 to 0.89]
Statistical Analysis 1: Comparison: Autopsy Cohort; Spearman's Rank Order Correlation of the median semiquantitative read (three readers) and the quantitative IHC measurement of cortical amyloid plaque density averaged across six brain regions; Test type: Superiority or Other; p < 0.0001, Spearman's Rank Correlation test — A one-sided test (rho > 0) was performed with a significance level of alpha=0.05 to assess a significant correlation; Correlation coefficient = 0.78, 95% CI 2-sided [0.58 to 0.89], Standard Error of Mean 0.194 — Asymptotic standard error and 95 percent CI used Fisher z-transformation

2. Primary Outcome: Specificity Analysis
Description: Specificity of florbetapir-PET scan in younger healthy controls presumed to be negative for amyloid. Specificity results are reported as the number of subjects who had a negative scan based on majority of 3 blinded readers.
Time Frame: 50-60 min after injection
Population: Per protocol, 27 subjects who were genetic carriers for ApoE e4 or whose genetic status was unknown were excluded from the analysis
Measure: Number; unit: participants
Arm/Group | Specificity Cohort
Number analyzed (Participants) | 47
participants
  Positive for amyloid | 0 [91 to 100]
  Negative for amyloid | 47
Statistical Analysis 1: Comparison: Specificity Cohort; Proportion of subjects who had a negative scan based on majority of 3 blinded readers; Test type: Superiority or Other; Specificity = 100, 95% CI 2-sided [91 to 100] — 95% CI calculated by Wilson score method

3. Secondary Outcome: Regional Correlation Analysis
Description: Spearman's rank order correlation of median visual read of the florbetapir-PET image vs. amyloid plaque density assessed post-mortem by quantitative IHC of six individual brain regions (precuneus, parietal cortex, frontal cortex, temporal cortex, posterior cingulate, anterior cingulate). Spearman's rank order correlation ranges from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: at autopsy up to 12 months post-scan
Population: All subjects with a valid image who came to autopsy within 1 year of scan, minus 6 subjects who served as front-runners
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 29
Correlation coefficient
  Precuneus | 0.75 [0.53 to 0.88]
  Parietal cortex | 0.77 [0.56 to 0.88]
  Frontal cortex | 0.69 [0.44 to 0.84]
  Temporal cortex | 0.68 [0.42 to 0.84]
  Posterior cingulate | 0.70 [0.44 to 0.85]
  Anterior cingulate | 0.74 [0.51 to 0.87]

ADVERSE EVENTS:
Time Frame: AEs were collected up to 48 hours after injection. SAEs were collected up to 30 days after injection.
Arm/Group | Autopsy Cohort | Specificity Cohort
Serious Adverse Events (participants affected / at risk) | 1/152 | 0/74
Other Adverse Events (participants affected / at risk) | 3/152 | 2/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autopsy Cohort (N=152) | Specificity Cohort (N=74)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (152) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autopsy Cohort (N=152) | Specificity Cohort (N=74)
Headache (Nervous system disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days